CLINICAL TRIAL: NCT01777308
Title: The Vaccine Response and Long-term Antibody Persistence of GSK Biologicals' MenACWY-TT Vaccine (GSK134612) Administered as One Dose at 6 Years Post-MenC Primary Vaccination in Healthy Subjects Aged 12-18 Months at Primary Vaccination
Brief Title: Immunogenicity, Reactogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' MenACWY-TT Vaccine Administered 6 Years Post-MenC Primary Vaccination in Healthy Subjects Who Were 12-18 Months at Primary Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116727; 2012-002575-34 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2017-09

CONDITIONS: Infections, Meningococcal
Keywords: Immunogenicity; Booster; Healthy; Vaccine response; Safety; Neisseria meningiditis; Antibody persistence; Meningococcal conjugate vaccine
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Menitorix Group (Experimental): Subjects who were primed with Menitorix™ (Hib-MenC-TT) + Priorix™ (MMR) vaccines in the primary study HIB-MENC-TT-016 (NCT00326118) received one dose of Nimenrix™ (MenACWY-TT) booster vaccine at Month 72 post primary vaccination (booster visit 1).
  The MenACWY-TT vaccine was administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Interventions: Biological: Meningococcal conjugate vaccine GSK134612
- Meningitec + Hiberix Group (Experimental): Subjects who were primed with Meningitec™ (MCC) + Hiberix™ (Hib) + Priorix™ (MMR) vaccine in the primary study HIB-MENC-TT-016 (NCT00326118) received one dose of Nimenrix™ (MenACWY-TT) booster vaccine at Month 72 post primary vaccination (booster visit 1).
  The MenACWY-TT vaccine was administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Interventions: Biological: Meningococcal conjugate vaccine GSK134612

INTERVENTIONS:
Biological: Meningococcal conjugate vaccine GSK134612 — Single dose to be administrated intramuscularly in the deltoid of the non-dominant arm

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, reactogenicity and safety of a booster dose of GSK Biologicals' MenACWY-TT vaccine administered at 6 years post-primary vaccination with either GSK Biologicals' Hib-MenC-TT vaccine (Menitorix™) or Hiberix™ and Meningitec™, in healthy subjects aged 12-18 months at primary vaccination and to evaluate the long-term antibody persistence at 2 years after MenACWY-TT booster vaccination.

This is an extension study of the Hib-MenC-TT-016 study (NCT number: NCT00326118).

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* A male or female between, and including, 84 and 95 months of age at the time of the booster vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject and written informed assent obtained from the subject in accordance with local laws and regulations.
* Healthy subjects as established by medical history and history-directed physical examination before entering into the study.
* Having completed the vaccination in the study [Hib-MenC-TT-016 (106445)] as per protocol.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after the study vaccine dose, with the exception of a licensed inactivated influenza vaccine which can be administered at any time during the study according to the local recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination with meningococcal vaccine except the meningococcal vaccination received in the Hib-MenC-TT-016 study.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including Human Immunodeficiency Virus (HIV)infection, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine, and history of serious allergic reaction (anaphylaxis) following the administration of vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures, including GBS. History of a simple, single febrile seizure is permitted.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the study vaccination or planned administration during the booster vaccination phase of the study (i.e. between Visit 1 and Visit 2) and within 3 months preceding the blood sampling at Visit 3.

The following criteria should be checked for the long-term persistence phase at two years after booster vaccination (Visit 3):

In case an exclusion criterion becomes applicable, the subject will not enter the long-term follow-up and the reason will be documented.

* Previous administration of a meningococcal vaccine with the exception of the meningococcal vaccination given in the primary study and the booster vaccination in this particular study.
* History of meningococcal disease.

Ages: 84 Months to 95 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2013-05-03; Primary Completion 2014-07-03 (Actual); Study Completion 2016-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Australia (8):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Subiaco, Western Australia

REFERENCES:
- [Derived] Nolan T, Booy R, Marshall HS, Richmond P, Nissen M, Ziegler JB, Baine Y, Traskine M, Jastorff A, Van der Wielen M. Immunogenicity and Safety of a Quadrivalent Meningococcal ACWY-tetanus Toxoid Conjugate Vaccine 6 Years After MenC Priming as Toddlers. Pediatr Infect Dis J. 2019 Jun;38(6):643-650. doi: 10.1097/INF.0000000000002334. PMID 31116180

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Menitorix Group: Healthy male or female subjects, who were primed with Menitorix vaccine (administered intramuscularly in the deltoid region of the left arm) and with Priorix vaccine (administered subcutaneously in the upper-right side of the arm) during the primary study HIB-MENC-TT-016 (NCT00326118), additionally received in the current study one booster dose of Nimenrix vaccine at Month 72 post-primary vaccination (Booster Visit 1). The Nimenrix vaccine was administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
- Meningitec + Hiberix Group: Healthy male or female subjects, who were primed with Meningitec vaccine (administered intramuscularly in the deltoid region of the non-dominant arm), with Hiberix vaccine (administered intramuscularly in the left side of the thigh) and with Priorix vaccine (administered subcutaneously in the upper-right side of the arm) during the primary study HIB-MENC-TT-016 (NCT00326118), additionally received in the current study one booster dose of Nimenrix vaccine at Month 72 post-primary vaccination (Booster Visit 1). The Nimenrix vaccine was administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Started | 119 | 37
Completed up to Month 73 | 118 | 37
Completed (Completed up to Month 96) | 105 | 34
Not Completed | 14 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Migrated/moved from study area | 1 | 0
Not completed — Lost to Follow-up | 7 | 2
Not completed — Blood draw refusal at Visit 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menitorix Group | Meningitec + Hiberix Group | Total
Number analyzed (Participants) | 119 | 37 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.0 (0.2) | 7.0 (0.0) | 7.0 (0.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 14 | 71
  Male | 62 | 23 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian-East Asian Heritage | 1 | 1 | 2
  Geographic ancestry: Asian-South East Asian Heritage | 1 | 0 | 1
  Geographic ancestry: White-Caucasian/European Heritage | 109 | 36 | 145
  Geographic ancestry: Asian - Central/South Asian Heritage | 1 | 0 | 1
  Geographic ancestry: Unspecified | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response for Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitides Serogroup A, C, W-135 and Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY)
Description: Vaccine response was defined as: For initially seronegative subjects (pre-vaccination rSBA titer below 1:8), antibody titer greater than or equal to (≥) 1:32 at post-vaccination; for initially seropositive subjects, antibody titer at post-vaccination ≥ 4 fold the pre-vaccination antibody titer.
Time Frame: At Month 73, one month post-booster vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Month 73, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month post-vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 104 | 34
Participants
  rSBA-MenA | 102 | 33
  rSBA-MenC | 101 | 33
  rSBA-MenW-135 | 102 | 33
  rSBA-MenY | 101 | 33

2. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ the Predefined Cut-off Values
Description: The cut-off values for the rSBA titers were greater than or equal to (≥) 1:8 and 1:128.
Time Frame: At Month 73, one month post-booster vaccination
Population: The analysis was performed on the Adapted ATP cohort at Month 73, which included all evaluable subjects from the ATP cohort for safety for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sample taken one month post-vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 104 | 35
Participants
  rSBA-MenA, ≥ 1:8 | 102 | 35
  rSBA-MenA, ≥ 1:128 | 102 | 35
  rSBA-MenC, ≥ 1:8 | 102 | 35
  rSBA-MenC, ≥ 1:128 | 102 | 34
  rSBA-MenW-135, ≥ 1:8 | 102 | 35
  rSBA-MenW-135, ≥ 1:128 | 102 | 35
  rSBA-MenY, ≥ 1:8 | 103 | 34
  rSBA-MenY, ≥ 1:128 | 103 | 34

3. Secondary Outcome: Antibody Titers Against rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 73, one month post-booster vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 104 | 35
Titer
  rSBA-MenA | 3421.4 [2659.3 to 4402] | 2925.1 [1949.5 to 4389]
  rSBA-MenC | 11819.2 [9026.4 to 15476.1] | 7419.7 [4543.2 to 12117.3]
  rSBA-MenW-135 | 17166.5 [12745.9 to 23120.3] | 15747.7 [10033 to 24717.7]
  rSBA-MenY | 4871 [3932.7 to 6033.1] | 3495.9 [2126.6 to 5746.8]

4. Secondary Outcome: Number of Subjects With Anti-tetanus (Anti-T) Concentrations ≥ the Predefined Cut-off Values
Description: The cut-off values for anti-T concentrations were greater than or equal to (≥) 0.1 international units per milliliter (IU/mL) and ≥ 1 IU/mL.
Time Frame: At Month 73, one month post-booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 103 | 34
Participants
  Anti-T ≥ 0.1 IU/mL | 103 | 34
  Anti-T ≥ 1 IU/mL | 102 | 33

5. Secondary Outcome: Antibody Concentrations Against Tetanus (Anti-T) Antigen
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL).
Time Frame: At Month 73, one month post-booster vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 103 | 34
IU/mL | 15.6 [13.1 to 18.6] | 12.5 [8.4 to 18.7]

6. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers ≥ the Predefined Cut-off Values
Description: The cut-off values for the rSBA titers were greater than or equal to (≥) 1:8 and 1:128.
Time Frame: At Month 96, 24 months post-booster vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for persistence at Month 96, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen at 24 months post booster vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 100 | 33
Participants
  rSBA-MenA, ≥ 1:8 | 72 | 21
  rSBA-MenA, ≥ 1:128 | 67 | 17
  rSBA-MenC, ≥ 1:8 | 100 | 31
  rSBA-MenC, ≥ 1:128 | 90 | 26
  rSBA-MenW-135, ≥ 1:8 | 96 | 30
  rSBA-MenW-135, ≥ 1:128 | 96 | 30
  rSBA-MenY, ≥ 1:8 | 95 | 29
  rSBA-MenY, ≥ 1:128 | 95 | 29

7. Secondary Outcome: Antibody Titers Against rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBa-MenY
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 96, 24 months post-booster vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 100 | 33
Titers
  rSBA-MenA | 174.9 [102.4 to 298.7] | 79.0 [29.6 to 210.4]
  rSBA-MenC | 333.1 [278.3 to 398.8] | 175.4 [104.1 to 295.5]
  rSBA-MenW-135 | 1002.9 [742.1 to 1355.5] | 941.5 [448.4 to 1976.9]
  rSBA-MenY | 929.3 [678.0 to 1273.7] | 512.0 [250.1 to 1048.3]

8. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms included pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-booster vaccination period at Month 72
Population: The analysis was performed on the Total Vaccinated cohort (TVc) for safety at Month 73, which included all vaccinated subjects in the study Hib-MenC-TT-016 (NCT00326118) with a Nimenrix™ booster vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 118 | 37
Participants
  Any Pain | 69 | 15
  Any Redness | 56 | 19
  Any Swelling | 30 | 8

9. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), headache, and fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-booster vaccination period at Month 72
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 118 | 37
Participants
  Any Fatigue | 31 | 10
  Any Gastrointestinal symptoms | 29 | 5
  Any Headache | 29 | 6
  Any Fever | 6 | 1

10. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period at Month 72
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 119 | 37
Participants | 0 | 0

11. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period at Month 72
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 119 | 37
Participants | 36 | 7

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period at Month 72
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 119 | 37
Participants | 0 | 0

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 12
Time Frame: From Month 72 up to study end, at Month 96
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
Number analyzed (Participants) | 119 | 37
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period; Solicited and unsolicited symptoms: during the 31-day (Days 0-30) post-vaccination period; SAEs: up to study end at Month 96.
Arm/Group | Menitorix Group | Meningitec + Hiberix Group
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/37
Other Adverse Events (participants affected / at risk) | 95/119 | 28/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menitorix Group (N=119) | Meningitec + Hiberix Group (N=37)
Erythema (Skin and subcutaneous tissue disorders) | 56 (56) | 19 (19)
Fatigue (General disorders) | 31 (31) | 10 (10)
Gastrointestinal disorder (Gastrointestinal disorders) | 29 (29) | 5 (5)
Headache (Nervous system disorders) | 30 (30) | 7 (9)
Pain (General disorders) | 69 (69) | 15 (15)
Pyrexia (General disorders) | 6 (6) | 2 (2)
Swelling (General disorders) | 30 (30) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.